CLINICAL TRIAL: NCT03062410
Title: Heath Related Quality of Life Assessment for Patients With Advanced or Metastatic Renal Cell Carcinoma Treated With Tyrosine Kinase Inhibitor Using Electronic Patient Reported Outcome in Daily Clinical Practice.
Brief Title: Quality of Life Assessment in Daily Clinical Oncology Practice for Patients With Advanced Renal Cell Carcinoma
Acronym: QUANARIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R/2016/54
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Renal Carcinoma Metastatic; Kidney Neoplasms; Renal Cancer
Keywords: Health Related Quality of Life; Routine clinical practice; Electronic Patient Reported Outcome; EORTC QLQ-C30; Pazopanib; Sunitinib; Tyrosine Kinase Inhibitor anti-VEGF; Patient Reported Outcome; Supportive Care; Quality of Life
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic PRO (Other): All patients diagnosed with mRCC initiating TKI anti-VEGF treatment (Sunitinib or Pazopanib) will be invited to complete the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 cancer specific questionnaire and the EQ-5D before each visit with the physician. Questionnaires completion will be done by patients on tablets and/or computer terminals via the CHES software (Computer-based Health Evaluation System) at hospital before consultation or at home via secured portal. Physician will immediately have access to a visual summary of HRQOL evaluation.
  Interventions: Other: Electronic PRO in daily clinical practice

INTERVENTIONS:
Other: Electronic PRO in daily clinical practice — All patients diagnosed with mRCC initiating TKI anti-VEGF treatment (Sunitinib or Pazopanib) will be invited to complete the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 cancer specific questionnaire and the EQ-5D before each visit with the physician. Questionnaires completion will be done by patients on tablets and/or computer terminals via the CHES software (Computer-based Health Evaluation System) at hospital before consultation or at home via secured portal. Physician will immediately have access to a visual summary of HRQOL evaluation.

SUMMARY:
Physician mainly use RECIST progression-free survival (PFS) and NCI CTCAE safety as a guide to evaluate treatment efficiency. In contrast Health Related Quality of Life (HRQOL) assessment is often restricted to clinical trial. It could be of particular interest to evaluate HRQOL in daily clinical practice in order to adequately choose and manage first line therapy, especially since HRQOL at diagnosis was shown to be a prognostic factor of overall survival in advanced or metastatic renal cell carcinoma (mRCC). A systematic collection in daily clinical practice of the HRQoL data using standardized questionnaires could strengthen management of symptoms : improve symptom control, improve patient-clinician communication, satisfaction with care and well-being of the patient and in fine the overall survival.

The objective of the QUANARIE Study is to assess the use of HRQOL assessment in daily clinical practice for patients with mRCC treated with tyrosine kinase inhibitor (TKI) using electronic patient reported outcome (PRO).

Indeed, the goal is to make the HRQoL data accessible and exploitable in real time to clinicians, to help medical professionals to optimize their practices by adopting a holistic and personalized approach based on patient reported outcomet.

DETAILED DESCRIPTION:
QUANARIE study is an interventional, prospective, multicenter trial involving 9 french oncological centers. Patients diagnosed with mRCC initiating TKI anti-VEGF treatment (Sunitinib or Pazopanib) will be invited to complete the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 cancer specific questionnaire and the EQ-5D before each visit with the physician. Questionnaires completion will be done by patients on tablets and/or computer terminals via the CHES software (Computer-based Health Evaluation System) at hospital before consultation or at home via secured portal. Physician will immediately have access to a visual summary of HRQOL evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal clear cells carcinoma, histologically or cytologically confirmed, locally advanced nonresectable or metastatic who initiate an oral treatment by ITK anti-VEGF (Pazopanib or Sunitinib.)
* Estimated life expectancy over than 3 months.
* Male or female
* Aged 18 years or older
* Patient able to understand French and to complete study questionnaires (no major cognitive disorders)
* Signed informed consent
* Patient affiliated to or beneficiary of French social security regime

Exclusion Criteria:

* Prior systemic treatment for metastatic renal cancer other than immunotherapy. Pretreatment or concomitant treatment with Biphosphonate or Denosumab is allowed.
* Renal carcinoma without clear cell component.
* Psychiatric illness compromising understanding of the information or conducting the study.
* Any acute or chronic disease (eg severe COPD) may affect the patient's ability to receive treatment under study or may make it difficult the interpretation of toxicities or adverse events.
* HIV positive.
* History of active chronic hepatitis including subjects who are carriers of Hepatitis B virus or Hepatitis C virus
* Uncontrolled infection
* History of digestive pathology which could compromise the good absorption of an oral ITK.
* Pregnancy, breast-feeding or absence/refusal of adequate contraception for fertile patients during the period of treatment and for 4 months from the last treatment administration.
* Hypersensitivity or contraindication to any of the study drugs (active substance of ITK or any excipients.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-11-04 (Estimated); Study Completion 2020-02-04 (Estimated)

PRIMARY OUTCOMES:
Rate of filled questionnaires at 12-months | 12 months
  Number of completed questionnaires compared to the number of consultations carried out during the first 12 months of follow-up.

SECONDARY OUTCOMES:
Exhaustiveness | 24 months
  Number of new cases for each center, initiating a treatment per ITK molecule compared to the number of patients to whom the intervention was proposed
Acceptability | 24 months
  Number of patients who agreed to participate in this study compared to the number of refusals on all patients, by center and by molecule type (Sunitinib or Pazopanib)
Effectiveness | 24 months
  Description of the toxicities collected by physicians according to the NCI CTCAE V4 compared to the toxicities reported by patients according to the 8 symptomatic dimensions of the QLC-C30 questionnaire and 9 items from EORTC Item Bank exploring 6 supplementary symptomatic dimensions
Physician satisfaction | 12 months

OTHER OUTCOMES:
Time to occurrence of grade 2 toxicity according to the NCI schedule CTCAE v4 | 24 months
  Defined as the time elapse between the inclusion date and the date of occurrence of grade 2 toxicity.
Survival under HRQoL deterioration | 24 months
  Assessed by the QLQ-C30 questionnaire and defined by the time between the inclusion date and the first clinically significant minimal deterioration (MCID) at the baseline score without clinically significant improvement or death from any cause
Time to treatment failure (TTF) | 24 months
  Defined as the time interval between the date of inclusion and death, tumor progression or definitive cessation of TKI treatment from any cause.
Progression-free survival (PFS): | 24 months
  Defined as the time interval between the date of inclusion and the date of first progression of the disease or death from any cause.
Overall Survival (OS): | 24 months
  Defined as the time interval between the date of inclusion and the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MOUILLET, MD, Principal Investigator — Centre Hospitalier Universitairede Besançon
Locations (8):
- France (8):
  - CHU de Besançon, Besançon
  - Hôpital privé Sainte Marie, Chalon-sur-Saône
  - Centre de lutte contre le cancer Georges François Leclerc, Dijon
  - Hôpital Nord Franche-Comté, Montbéliard
  - Centre de lutte contre le cancer Jean Godinot, Reims
  - Groupe hospitaliser St-Vincent, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre de lutte contre le cancer Alexis Vautrin - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mouillet G, Fritzsch J, Paget-Bailly S, Pozet A, Es-Saad I, Meurisse A, Vernerey D, Mouyabi K, Berthod D, Bonnetain F, Anota A, Thiery-Vuillemin A. Health-related quality of life assessment for patients with advanced or metastatic renal cell carcinoma treated with a tyrosine kinase inhibitor using electronic patient-reported outcomes in daily clinical practice (QUANARIE trial): study protocol. Health Qual Life Outcomes. 2019 Feb 4;17(1):25. doi: 10.1186/s12955-019-1085-1. PMID 30717745